CLINICAL TRIAL: NCT02128802
Title: Weight Reduction Surgery Followed by Kidney Transplantation for Patients With Class III Obesity and Renal Failure
Brief Title: Obesity Surgery and Kidney Transplant for Patients With Obesity and Renal Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Seth Karp, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130912
Record Dates: First submitted 2014-04-23; First posted 2014-05-01 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Severe Obesity; Renal Failure
Keywords: Obesity; Renal failure; Gastric bypass
MeSH Terms: conditions — Obesity, Morbid; Renal Insufficiency; Obesity | interventions — Gastric Bypass; Weight Reduction Programs

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical Gastric Bypass (Experimental): Patients will undergo surgical gastric bypass according to standard institutional protocols
  Interventions: Procedure: Gastric Bypass
- Medical Weight Loss Management (Experimental): Patients will receive best practices medical management for weight loss under current institutional protocols
  Interventions: Other: Weight Loss Program

INTERVENTIONS:
Procedure: Gastric Bypass
  Arms: Surgical Gastric Bypass
Other: Weight Loss Program
  Arms: Medical Weight Loss Management

SUMMARY:
Gastric Bypass followed by renal transplantation is superior to medical management followed by renal transplant for patients with severe obesity and renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 40-55 kg/m2
* Age less than 60 years
* Available support person
* Adequate insurance
* All other criteria required for renal transplantation

Exclusion Criteria:

* Schizophrenia
* Bipolar disorder
* Crohn's disease
* Human Immunodeficiency Virus
* Cirrhosis
* Prior weight loss surgery
* Prior mesh hernia repair
* Prior anti-reflux surgery
* Inability to walk 200 feet
* Significant coronary disease
* Significant lung disease - Fixed expiratory volume 1 less than 75% or on oxygen
* Addiction to alcohol or drugs
* Inability to quit smoking
* Jehovah's witness
* Non-compliance with dialysis regimen
* Previous renal transplant
* Non-English speaking

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Ability to reach medical suitability for renal transplant within 18 months after initiating treatment and the change and trajectory of health-related quality of life (HRQOL) | 18 months
  Outcomes will be measured based on weight loss and a variety of validated surveys and questionnaires to measure HRQOL

SECONDARY OUTCOMES:
All-cause mortality | 5 years
  Number of patients who die from any cause
Weight loss | 5 years
  Amount of weight lost at various points over the study period
Surgical outcomes | 5 years
  Incidence of surgical complications including but not limited to leak rate, stricture rate, pulmonary embolism, and infection.
Development or regression of diabetes | 5 years
  Including but not limited to start of stop of insulin therapy, amount of insulin required, and start or stop of or cal medications.
Development or regression of other comorbidities | 5 years
  Development or regression of other diseases including but not limited to hypertension, coronary artery disease, and skin infections.
Health care utilization | 5 years
  This outcome measure includes but is not limited to the amount of money spent on health care, total hospitalization, days of hospitalization, and procedures required.
Nutritional status | 5 years
  This outcome includes but is not limited to measures of albumin, pre-albumin, and caloric intake.
Hormonal and metabolic status | 5 years
  This outcome includes but is not limited to measurement of protein catabolism, creatinine clearance, and serum prealbumin. In addition, protein and iron metabolism will be measured using serum albumin, transferrin and ferritin. Glucose metabolism will be measured by glucose and insulin levels. regression of the disease. Lipid metabolism will be assessed with triglyceride levels, very-low density lipoproteins, and cholesterol. Micronutrient levels will be measured with vitamin D, thiamin, B12, and folate.

OTHER OUTCOMES:
Prograf dosing | 5 years
  This outcome will assess the amount of prograf required for therapeutic levels

CONTACTS AND LOCATIONS:
Overall Officials: Seth Karp, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States